CLINICAL TRIAL: NCT01073579
Title: Sabril Patient Registry
Status: Completed | Type: Observational
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13101A; OV1040 (Other: Former study ID)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Infantile Spasms; Refractory Complex Partial Seizures in Adults
Keywords: Cryptogenic Infantile Spasms; Cryptogenic West Syndrome; Hypsarrhythmia; Infantile Spasms; Symptomatic Infantile Spasms; Symptomatic West Syndrome; West Syndrome; Refractory Complex Partial Seizures; Complex Partial Epilepsy; Complex Partial Seizure Disorder; Cryptogenic Partial Complex Epilepsy; Disorder, Complex Partial Seizures; Epilepsy, Cryptogenic, Partial Complex; Epilepsy, Psychic Equivalent; Epilepsy, Psychomotor; Epilepsy, Symptomatic, Partial Complex; Partial Complex Epilepsy, Cryptogenic; Partial Complex Epilepsy, Symptomatic; Seizure Disorder, Complex Partial; Symptomatic Partial Complex Epilepsy
MeSH Terms: conditions — Spasms, Infantile; Seizures; Epilepsy, Complex Partial | interventions — Vigabatrin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sabril®: All patients in the U.S. who are prescribed Sabril must participate in this patient registry in order to receive Sabril.
  Interventions: Drug: Sabril®

INTERVENTIONS:
Drug: Sabril® — Infantile Spasms (IS): Initiate therapy at 50 mg/kg/day twice daily increasing total daily dose per instructions to a maximum of 150 mg/kg/day.
  Refractory Complex Partial Seizures (rCPS) in Adults: Initiate therapy at 500 mg twice daily, increasing total daily dose per instructions. The recommended dose is 1.5 grams twice daily.
  Other Names: Vigabatrin

SUMMARY:
The purpose of this study is to create a patient registry to collect and analyze information on subjects treated with Sabril and the prescribers of Sabril.

DETAILED DESCRIPTION:
This prospective registry is part of the overall Risk Evaluation and Mitigation Strategy (REMS) required for Sabril by the United States Food and Drug Administration (FDA). All physicians who prescribe Sabril and all patients who take Sabril will be enrolled in a H. Lundbeck A/S-sponsored program called "SHARE" (Support, Help and Resources for Epilepsy), and the data that are collected and entered into the SHARE database will form the basis of this patient registry.

Prior to any prescription being filled by one of the specialty pharmacies, the prescribing physician and the patient must be enrolled in SHARE. A call center (SHARE Call Center) will act as the hub for a network of select specialty pharmacies. Participation in both SHARE and the patient registry is mandatory.

Information regarding prescriber specialty and location, patient demographic and disease characteristics will be collected through SHARE and entered into the database. Patients will be assigned a unique patient identifier upon entry into the registry, and all data related to that patient will be associated with this identifier.

Early in therapy (within 2-4 weeks for Infantile Spasms patients and 3 months for adult refractory Complex Partial Seizures patients), a mandatory benefit/risk assessment will occur. If the benefit of Sabril therapy exceeds the risk of vision loss, the prescribing physician will complete and submit the appropriate SHARE form and the patient will continue into the maintenance therapy phase of treatment. The outcome of this benefit/risk assessment will be entered into the database.

Regular assessments of vision are required during Sabril therapy to contribute information related to the ongoing benefit/risk assessments. The required assessments will occur at baseline, every 3 months during therapy, and about 3-6 months after stopping Sabril. The visual assessment results will be recorded and submitted using the appropriate SHARE forms, and the data will be entered into the database. A copy of the visual field will be included.

Patients will participate in the registry for as long as they receive Sabril therapy. Patients who discontinue treatment with Sabril, but are treated with it again at a later time will be treated as a single patient in the registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the U.S. who are prescribed Sabril must participate in this patient registry in order to receive Sabril.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the U.S. who are prescribed Sabril must participate in this patient registry in order to receive Sabril. There are no other eligibility criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 9423 (Actual)
Dates: Start 2009-08; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Characterize the prevalence, incidence, time to onset, progression, and severity of vision loss during Sabril treatment. | A yearly report

SECONDARY OUTCOMES:
Characterize the demographics, disease characteristics, dose and duration of therapy for patients who receive Sabril. | A yearly report
Characterize the physician specialties for prescribers of Sabril. | A yearly report

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com